CLINICAL TRIAL: NCT00002848
Title: SUPPORTIVE-EXPRESSIVE GROUP THERAPY FOR MEN WITH PRIMARY PROSTATE CANCER
Brief Title: Group Therapy Compared With Educational Materials in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC CCOP Research Base, University of Rochester
Organization: University of Rochester (Other)
Other Study IDs: CDR0000065087; URCC-U9994; NCI-CCC-94-32; URCC-9994P(A); NCI-P96-0072
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Developing coping strategies may help improve the quality of life of patients with prostate cancer.

PURPOSE: This randomized clinical trial is comparing the effect of group therapy with written educational materials on the quality of life of men with stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of providing group support, and evaluate the effect of supportive-expressive group therapy vs. written educational material on the psychological health and quality of life of men with stage I/II prostate cancer.

OUTLINE: Patients are stratified by prior hormonal therapy.

Patients continue standard oncologic treatment concurrently with supportive-expressive group therapy.

Supportive-expressive group therapy consists of twelve 90-minute weekly meetings with 8-12 members and 2 cotherapists and is based on the following themes: building bonds, expressing emotions, detoxifying dying, taking time to prioritize and set realistic goals, fortifying families, and dealing with doctors. Each session commences with a brief stress reduction exercise and ends with a brief cognitive restructuring imagery exercise. The main portion of the meeting emphasizes providing an environment in which patients can share their concerns, feelings, and thoughts openly and honestly. The role of the cotherapist is to facilitate expression of patients' concerns, offer empathy, and continue to encourage patients to express their feelings and thoughts.

Quality-of-life questionnaires are filled out at 3 and 6 months and then every 6 months for a total of 2 years.

PROJECTED ACCRUAL: Approximately 480 patients (including an estimated 53 minority patients) will be entered in this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven prostate cancer diagnosed within 1 year prior to entry

  * Clinical stage I/II (T1b-c or T2, N0 or Nx, M0) disease

    * Pathologic local upstaging (e.g., to T3) allowed

      * No Nx disease if pathologic or partial pathologic (e.g., lymph node biopsy or dissection) staging performed
* No major psychiatric illness requiring hospitalization or medication other than depression or anxiety for less than 1 year
* No second malignancy within 10 years except nonmelanomatous skin cancer
* Clinical follow-up by a urologist, medical oncologist, or radiation therapist required at least semi-annually

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 1997-04; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, PhD, MS, Study Chair — James P. Wilmot Cancer Center
Locations (7):
- United States (7):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Northwest, Tacoma, Washington